CLINICAL TRIAL: NCT06138847
Title: Does Levetiracetam and Carbamazepine Impact the Autonomic Activity of Children With Self-limiting Focal Epilepsy?
Acronym: levcbz
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: İpek Dokurel (Other)
Responsible Party: Sponsor-Investigator, İpek Dokurel, İpek Dokurel Çetin,MD, Ege University
Organization: Ege University (Other)
Other Study IDs: levcbzepilepsy
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy; Syndrome, Seizures of Localized Onset
Keywords: Heart rate variability; epilepsy; children; carbamazepine; levetiracetam; rSUDEP-7
MeSH Terms: conditions — Epilepsy; Syndrome | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Group I consisted of children with epilepsy who were only taking one type of ASMs, either levetiracetam or carbamazepine
  Interventions: Diagnostic Test: electroencephalogram
- Group II: Group II comprised forty-one age and sex-matched healthy children as a control group.

INTERVENTIONS:
Diagnostic Test: electroencephalogram — Polygraphic derivations generally include an ECG channel, which is standard on EEG recordings, plus an optional EMG channel. Subsequently, the signal was recorded at 512 Hz and inspected using the standard bipolar and referential montages
  Groups: Group I

SUMMARY:
The goal of this cross-sectional study is to learn about autonomic cardiac profile changes in children with self-limiting focal epilepsy using levetiracetam and carbamazepine in children with self-limiting focal epilepsy syndrome. The main questions is it aims to answer are:

1. Are heart rate variability and autonomic tone different among healthy controls and children with epilepsy?
2. Does Levetiracetam and carbamazepine affect autonomic tone differently among children with self-limiting focal epilepsy?

DETAILED DESCRIPTION:
Seventy-eight children with self-limiting focal epilepsy syndrome were enrolled in the study and were divided into two groups. Group I consisted of children with epilepsy who were only taking one type of ASM, either levetiracetam or carbamazepine. They were further subdivided into group Ia, which included patients receiving levetiracetam, and group Ib, which included patients receiving carbamazepine. Group II comprised forty-one age and sex-matched healthy children as a control group.

The pediatric neurologist utilized the clinical definition criteria of the International League Against Epilepsy to diagnose all children with self-limiting focal epilepsy syndrome.

The demographics, clinical data, neuroimaging findings, interictal scalp EEG results, and outcomes of patients' medical records were examined retrospectively. Utilizing the 10-20 system, gold cup electrodes (accompanied by conductive paste and collodium) were placed and used to acquire scalp recordings. Polygraphic derivations generally include an ECG channel, standard EEG recordings, plus an optional EMG channel.

All subjects had echocardiographic (ECHO) testing using M-mode, 2-dimensional, color, pulse, and continuous wave Doppler echocardiograms with a GE Vivid S6. A standard ambulatory electrocardiography (ECG) recording system (Cardioline Click Holter HRV Package System, version 1.4.1 Biomedical Systems, Italy) was used. All of the patients were examined during an at least 24- hour seizure-free period, and none of the patients reported seizures during the recording period and encouraged to perform their normal daily activities. Artifacts and ectopic complexes were excluded. Heart rate variability parameters used for the time domain analysis were the mean and the highest and lowest heart rates. Time domain analysis included the following: standard deviation (SD) of all normal RR intervals (SDNN, ms), SD of the average normal sinus intervals between successive heartbeats (RR intervals) for all 5 min segments of the entire recording (SDANN, ms), the root mean squares successive differences RR intervals (RMSSD, ms), the proportion of the adjacent RR intervals that differ by more than 50 ms in the 24- hour recording (pNN50, measured in percentage). While the RMSSD and pNN50 reflect vagally mediated (i.e., parasympathetic) HRV, the SDNN represents the parasympathetic and sympathetic components of the autonomic nervous system.

The rSUDEP-7 inventory was used to assess group I risk for SUDEP. The SUDEP-7 was found to be associated with a biomarker of vagus-mediated HRV(RMSSD)[25]. The revised SUDEP-7 Risk Inventory incorporates seven validated risk factors (Table 1). Since our study cohort consisted of the pediatric age group and the study design was based on patients receiving monotherapy, none of group 1 received points from the 5th and 6th items of the risk factor list.

ELIGIBILITY:
Inclusion Criteria:

* Based on the ILAE classification, all children with epilepsy are categorized as self-limiting focal epilepsy syndromes.

Exclusion Criteria:

* had signs of organic heart disease
* had other conditions that could influence the cardiovascular and autonomic nervous systems (such as systemic lupus erythematosus, and endocrine-metabolic abnormalities)
* use regular medications that have an impact on the cardiovascular and autonomic nervous systems

Ages: 5 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Seventy-eight children aged 5-17 years old with with self-limiting focal epilepsy syndrome were enrolled in the study and were divided into two groups. Group I consisted of children with epilepsy who were only taking one type of ASMs, either levetiracetam or carbamazepine. They were further subdivided into group Ia, which included patients receiving levetiracetam and group Ib, which included patients receiving carbamazepine. Group II comprised forty-one age and sex-matched healthy children as a control group.
Sampling Method: Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
children with epilepsy has autonomic disfunction | 1-5 months
  children with self-limiting focal epilepsy syndrome on monotherapy evinced parasympathetic cardiac autonomic dysfunction when measured by time domain heart rate variability as opposed to healthy individuals

CONTACTS AND LOCATIONS:
Overall Officials: Muhlike Guler, MD, Study Director — Balikesir Ataturk City Hospital
Locations (1):
- Balıkesir University Medical Faculty, Merkez, Balikesi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hennessy MJ, Tighe MG, Binnie CD, Nashef L. Sudden withdrawal of carbamazepine increases cardiac sympathetic activity in sleep. Neurology. 2001 Nov 13;57(9):1650-4. doi: 10.1212/wnl.57.9.1650. PMID 11706106
- [Background] Mukherjee S, Tripathi M, Chandra PS, Yadav R, Choudhary N, Sagar R, Bhore R, Pandey RM, Deepak KK. Cardiovascular autonomic functions in well-controlled and intractable partial epilepsies. Epilepsy Res. 2009 Aug;85(2-3):261-9. doi: 10.1016/j.eplepsyres.2009.03.021. Epub 2009 May 5. PMID 19409754